CLINICAL TRIAL: NCT01719913
Title: Gut, Grain and Greens (3G): The Effect of Gluten on Gut Microbiome and Metabolic Health.
Brief Title: The Effect of Gluten on Gut Microbiome and Metabolic Health.
Acronym: 3G
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Oluf Borbye Pedersen, Scientific Director, professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NNF-CBMR 3861-34275
Record Dates: First submitted 2012-10-24; First posted 2012-11-01 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Metabolic Diseases; Injury of Gastrointestinal Tract
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low gluten (Active Comparator): Poor gluten diet: Participants consume less than 5g gluten per day (estimated to correspond to a gluten intake below the 10th percentile in the population)
  Interventions: Other: Low gluten
- High gluten (Placebo Comparator): Refined grain/ gluten rich diet : Participants consume more than 25g of gluten per day (estimated to correspond to a gluten intake around the 90th percentile in the population)
  Interventions: Other: High gluten

INTERVENTIONS:
Other: High gluten — Refined grain/ gluten rich diet : Participants consume more than 25g of gluten per day (estimated to correspond to a gluten intake around the 90th percentile in the population)
  Arms: High gluten
Other: Low gluten — Poor gluten diet: Participants consume less than 5g gluten per day (estimated to correspond to a gluten intake below the 10th percentile in the population)
  Arms: Low gluten

SUMMARY:
Objective: To identify how specific changes of the gluten content in the diet affect the host-gut microbiome interactions with implications for metabolic health.

Design: A randomized, controlled, single-blinded, cross-over intervention trial consisting of two 8-week interventions periods, separated by a 6-week wash-out period. A total number of 60 participants will be included.

Intervention: low vs high gluten intake.

DETAILED DESCRIPTION:
The study is designed as a randomized, controlled, single-blinded, cross-over intervention trial consisting of two 8-week interventions periods, separated by a 6-week wash-out period. A total number of 60 participants will be included. Participants consume, in randomized order, a gluten-poor diet (<5 g/d) in the active treatment period and a gluten-rich diet (>25 g/d) during the control period.

Measurements: Altered quantitative metagenomics at bacterial gene- and species levels is the primary outcome of this study. Secondary outcomes include metabolic and inflammatory markers, circulating appetite hormone levels,serum metabolomics, gastrointestinal transit time and intestinal permeability. Furthermore, selected control measures are included; 4-day food records and a study intervention dietary records.

ELIGIBILITY:
Inclusion Criteria, compulsory:

* Body mass index (BMI): 25 - 35 kg/m2 OR
* Abdominal obesity: waist circumference: men: ≥ 94cm; women: ≥ 80cm
* No medically prescribed diet
* Weight stable
* Intense sporting activities less than 10 h/week
* Alcohol consumption less than 14 units/week (female) and 21 units/week (male)
* Signed informed consent

Inclusion criteria, minimum one of the following:

* Fasting plasma glucose from 6.1 mmol/l to 6.9 mmol/l
* Reduced high density lipoprotein (HDL) cholesterol; HDL ≤ 1.03 mmol/L for men and ≤ 1.29 mmol/L for women
* Increased triglyceride (TG) > 1.3 mmol/L
* Systolic blood pressure > 130 mmHg

Exclusion Criteria:

* Pharmacological treatment; diabetes and blood lipid regulation
* Lactating (or lactating, 6 weeks ago), pregnant (or pregnant, 3 months ago) or wish to become pregnant during the study
* Participation in another biomedical trial 1 month prior to study start
* Diagnosed with any form of diabetes, celiac disease or chronic pancreatitis
* Reported chronic gastrointestinal disorders
* Antibiotic treatment for 3 month prior to study start
* Blood hemoglobin < 7.0 mmol/l
* Blood donation within 1 month prior to study start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Altered quantitative metagenomics at bacterial gene- and species levels. | Up to 3 years.
  Feces samples are collected according to standard operation procedures for subsequent standardized microbial DNA extraction. Microbial DNA will be subjected to sequencing, microbial gene analyses, taxonomy analyses including enterotypes known species and unknown meta-species and functional annotation.

SECONDARY OUTCOMES:
Mean intestinal transit time | Up to 2 years.
  Participants are instructed in swallowing capsules containing different small non-invasive and non-absorbable plastic pellets for 6 consecutive days. On the seventh day they are having an X-ray of the abdomen taken.
Gastrointestinal permeability. | Up to 2 years.
  Lactulose/mannitol ratio in urine after four hours collection following oral intake of lactulose and mannitol.
Colonic fermentation | Up to 2 years.
  Breath hydrogen after intake of standardized breakfast (30,60,90,120,180 minutes)
Blood pressure and pulse. | Up to 1 year.
  Systolic and diastolic blood pressure and heart beat rate are measured after 10 min of rest according to current standard operational procedure with an automatic blood pressure meter. Participants are instructed not to talk during the measurements.
Saliva microbial flora | Up to 2 years.
  Saliva is collected after the participants have taken a small piece of paraffin in their mouth and have chewed until the paraffin has turned into one coherent mass (approximately one minute). Participants are swallowing the produced saliva for that minute. After this, and for the next 3 minutes, saliva is collected in a cup and handed over to the study personnel. Saliva is stored at minus 80 degrees for later studies of saliva microbial flora and saliva biochemistry.
Nasal fluid | Up to 3 years.
  Nasal fluid is collected by a non-invasive methodology for in vivo measurement of an array of immunological signalling molecules in the nasal airway lining. The method is based on a standardized collection of mucosal airway fluid from both nostrils onto small sheets of filter papers with efficient absorption properties. The technique is highly reproducible, and used for measuring immunological mediators representing the immediate response ability of the mucosal immune system.
Appetite hormones | Up to 3 years.
  Glucagon like peptide 1 and 2, Gastric inhibitory polypeptide, peptide YY and Ghrelin.
Celiac disease markers | Up to 1 year.
  Levels of gliadin and Immunoglobulin A and G transglutaminase.
Blood lipid profile | Up to 2 years.
  Low density Lipoproteins, High density lipoproteins, Total Cholesterol, Very low density lipoproteins and Free fatty acids.
Bioimpedance | Up to 1 year.
  Body composition (lean body mass and fat mass) is measured by bio-electrical impedance using multi frequency Quadscan.
Breath hydrogen. | Up to 2 years.
  Breath hydrogen measurements are done before the intake of the standardized breakfast (at 30, 60, 90, 120, 180 minutes), as an indicator of colonic fermentation.
Insulin | Up to 2 years.
  Fasting insulin and post prandial at 30, 60, 90, 120 and 180 minutes after standardized meal.
Glucose | Up to 2 years.
  Fasting glucose and post prandial at 30, 60, 90, 120 and 180 minutes after standardized meal.
C-peptide | Up to 2 years.
  Fasting.
Inflammatory makers | Up to 3 years.
  High sensitive C-reactive protein, Interleukin 1, 6 and 10, Lipopolysaccharide- binding protein, Tumor necrosis factor - alfa.
Anthropometric characteristics. | Up to 1 year.
  Weight, height, sagittal height and waist circumference.

OTHER OUTCOMES:
4 days precoded food diary. | Up to 2 years.
  Validated method for dietary registration, based on 2 week and 2 weekend days.
Gastrointestinal symptoms. | Up to 2 years.
  Changes from baseline to after intervention in individual gastrointestinal symptoms by validated VAS-questionary.

CONTACTS AND LOCATIONS:
Overall Officials: Oluf B Pedersen, MD, DMSCi,Professor, Principal Investigator — University of Copenhagen
Locations (1):
- The Novo Nordisk Foundation of Basic Metabolic Health, Section for Metabolic Genetics, Copenhagen, Denmark

REFERENCES:
- [Derived] Lind MV, Lauritzen L, Vestergaard H, Hansen T, Pedersen O, Kristensen M, Ross AB. One-carbon metabolism markers are associated with cardiometabolic risk factors. Nutr Metab Cardiovasc Dis. 2018 Apr;28(4):402-410. doi: 10.1016/j.numecd.2018.01.005. Epub 2018 Jan 31. PMID 29499850
- See also: Related Info — http://www.3g-center.dk/